CLINICAL TRIAL: NCT00611871
Title: The Use of Propranolol to Block Memory Reconsolidation in Post Traumatic Stress Disorders (PTSD)
Brief Title: The Use of Propranolol to Block Memory Reconsolidation in PTSD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment, grant term expired
Sponsor: Wayne State University (Other)
Collaborators: John D. Dingell VA Medical Center (U.S. Federal Agency); New York University (Other)
Responsible Party: Principal Investigator, Deane Aikins, Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HIC 0703002443
Record Dates: First submitted 2008-01-01; First posted 2008-02-11 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Posttraumatic Stress Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Propranolol following traumatic memory
  Interventions: Drug: Propranolol
- 2 (Active Comparator): Propranolol following neutral memory
  Interventions: Drug: Propranolol
- 3 (Placebo Comparator): Placebo following traumatic memory
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — 40mg propranolol, followed 2 hrs after with 60mg propranolol, immediately following memory recollection
  Arms: 1; 2
Drug: Placebo — 40mg placebo, followed 2 hrs after with 60mg placebo
  Arms: 3

SUMMARY:
The purpose of this investigation is to see if propranolol will reduce the psychophysiological hyperactivation associated with memories of combat stress in Veterans with Posttraumatic Stress Disorder.

DETAILED DESCRIPTION:
The goal of this translational research project is to generate a pilot sample of data from an investigation of a novel therapeutic approach to post traumatic stress disorder (PTSD). Current treatments for PTSD include exposure and other aspects of cognitive therapy as well as drug therapies based on serotonin-reuptake inhibiting antidepressant agents. However, these treatments are often unsuccessful, and symptoms in affected individuals may persist for decades. The central hypothesis guiding this research project posits that acquired fear responses, such as those in PTSD, when reactivated by recall become sensitive to noradrenergic modulation and thus may be permanently attenuated by blocking noradrenergic transmission. Further, we predict that this attenuation will facilitate subsequent therapy. In the current study, we will be investigating this model in three groups of Veterans of either Operation Iraqi Freedom or Operation Enduring Freedom (OIF/OEF) with PTSD: 1) Individuals who receive propranolol following recall of a traumatic memory (Propranolol-trauma); 2) Individuals who receive a placebo following recall of a traumatic memory (Placebo-trauma), and; 3) Individuals who receive propranolol following recall of an affective neutral memory (Propranolol-neutral). In addition, traumatic memory recall will be psychophysiologically assessed by measuring Veterans' facial corrugator electromyography (EMG), skin conductance, blood pressure and cardiovascular inter-beat interval responses pre- and one month post-medication administration.

ELIGIBILITY:
Inclusion Criteria:

* Participants will meet the clinical criteria of PTSD (DSM IVTR) secondary to combat exposure.

Exclusion Criteria:

* Current illicit substance use or alcohol consumption, as determined by urine toxicology and alcohol breath test.
* Any diagnosis of current comorbid psychotic disorders, bipolar disorder, or illicit substance or alcohol abuse or dependence.
* Any current prescription medication usage or supplement (dietary or herbal) usage that is contraindicated with propranolol.
* Active enrollment into any psychiatric or psychological treatment.
* Any condition that contraindicates the use of propranolol, such as:

  * history of bronchial asthma.
  * heart block.
  * sinus bradycardia.
  * congestive heart failure.
  * insulin-dependent diabetes.
  * initial systolic blood pressure < 100 mmHg.
  * Hyperthyroidism.
  * Thyroid disease.
  * Renal or liver impairment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-09; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Facial corrugator EMG | Change in Facial corrugator EMG from baseline at 1 month post-intervention

SECONDARY OUTCOMES:
CAPS score | Change in CAPS score from baseline at 1 month post-intervention
PCL-M score | Change in PCL-M score from baseline at 1 month post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Deane Aikins, PhD, Principal Investigator — Wayne State University
Locations (1):
- John D Dingell VA Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No